CLINICAL TRIAL: NCT03834441
Title: Optimized Health-Related Social Needs Screening and Community Linkages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Margaret Samuels-Kalow, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019P000128
Record Dates: First submitted 2019-02-05; First posted 2019-02-08 (Actual); Results first posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Emergencies
Keywords: social needs
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral screening (Other)
  Interventions: Other: Oral HRSN screening
- Written screening (Other)
  Interventions: Other: Written HRSN screening

INTERVENTIONS:
Other: Oral HRSN screening — Verbal screening delivered by an RA
  Arms: Oral screening
Other: Written HRSN screening — Patient completes written screen on iPad.
  Arms: Written screening

SUMMARY:
The objective of this study is to to understand the most effective method for health-related social need (HRSN) screening in the challenging environment of an emergency department by randomizing patients to oral or written HRSN screening in the ED.

DETAILED DESCRIPTION:
Bilingual research assistants (RA) will screen patients for eligibility based on the predetermined criteria and approach eligible patients with a brief description of the study and opportunity for participation. Interested participants will complete a verbal consent process to reduce the barriers to participation, a brief demographic questionnaire, and an assessment of health literacy (Newest Vital Sign) followed by the Partners Healthcare HRSN screener randomized to an oral v. iPad screening strategy.

After completion of the screening tool, participants will complete a secondary questionnaire asking about satisfaction with the process, the presence of additional HRSN not recorded by the Partners HealthCare screener, and their perspectives on screening. At the conclusion, all participants will be provided with standardized, bilingual list of community resources to address each of the screening domains.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years patients and either a parent/guardian of a pediatric/cognitively disabled patient in the MGH ED,
2. triaged to the Acute, CDU, Fast Track, Urgent, and Pediatrics areas,
3. English- or Spanish-speaking, and
4. capable of informed consent.

Exclusion Criteria:

1. patients unwilling to have the interview audio-recorded,
2. medically unstable patients, and
3. Section 12, lack of capacity medical hold, sexual assault, child abuse, and emotionally distressed patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Samuels-Kalow, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

RESULTS

PARTICIPANT FLOW:
Period: Allocation
Arm/Group | Oral Screening | Written Screening
Started | 115 | 121
Completed | 112 | 116
Not Completed | 3 | 5
Period: Analysis
Arm/Group | Oral Screening | Written Screening
Started | 112 | 116
Completed | 105 | 109
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Screening | Written Screening | Total
Number analyzed (Participants) | 115 | 121 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (15) | 39 (15) | 40 (15)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 42 | 55 | 97
  Female | 72 | 64 | 136
  Other | 0 | 1 | 1
  Missing | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 25 | 28 | 53
  White NH | 65 | 72 | 137
  Black NH | 9 | 5 | 14
  Other NH | 14 | 16 | 30
  Missing/declined | 2 | 0 | 2
Health literacy [Number; unit: participants]
  Adequate | 69 | 72 | 141
  Limited | 42 | 46 | 88
  Missing | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Satisfaction With the Screening Process
Description: Satisfaction with screening as measured by:
  Please tell us how satisfied you were with the questionnaire you just took:
  Extremely Quite a bit Somewhat A little bit Not at all
Time Frame: Immediately after completing survey
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Screening | Written Screening
Number analyzed (Participants) | 115 | 121
Participants
  Extremely/quite a bit | 94 | 97
  Somewhat/a little/ not at all | 12 | 15
  Missing | 9 | 9

2. Secondary Outcome: Number of Health Related Social Needs Reported
Description: We will record the number of health related social needs reported
Time Frame: Immediately after completing survey
Population: Would you like any information about any of the HRSN topics?
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Screening | Written Screening
Number analyzed (Participants) | 115 | 121
Participants
  None | 70 | 93
  At least one | 45 | 28

ADVERSE EVENTS:
Time Frame: Through study completion (no more than 1 day).
Description: Participants were enrolled in the study and completed the outcome measurement on the same day. There was no further contact with participants.
Arm/Group | Oral Screening | Written Screening
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/121
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/121
Other Adverse Events (participants affected / at risk) | 0/115 | 0/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT03834441/Prot_000.pdf